CLINICAL TRIAL: NCT01078779
Title: A Randomised, Double-blind, Placebo Controlled Trial of Chloroquine for the Prevention of Influenza
Brief Title: The Chloroquine for Influenza Prevention Trial
Acronym: CHIP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Professor Nicholas Paton, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: E/09/482
Record Dates: First submitted 2010-02-28; First posted 2010-03-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Influenza
Keywords: Influenza; Prevention; Chloroquine; Randomised controlled trial; Respiratory virus infection
MeSH Terms: conditions — Influenza, Human | interventions — Chloroquine; chloroquine diphosphate; Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chloroquine (Experimental)
  Interventions: Drug: Chloroquine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chloroquine — Chloroquine phosphate 250mg capsule, two capsules daily for 7 days then 2 capsules once a week for a total treatment duration of 12 weeks
  Other Names: Chloroquine phosphate; Plaquenil
  Arms: Chloroquine
Drug: Placebo — Placebo capsules, 2 capsules daily for 7 days then 2 capsules weekly for a total treatment duration of 12 weeks
  Arms: Placebo

SUMMARY:
A randomised controlled trial to determine the efficacy of chloroquine for the prevention of influenza

ELIGIBILITY:
Inclusion Criteria:

* Age 18 -65
* Have the ability to provide informed consent
* If a woman of child-bearing potential, willing to use contraception for the period of the trial

Exclusion Criteria:

* Acute influenza-like illness at screening
* History of psoriasis, porphyria cutanea tarda, epilepsy, myasthenia gravis, myopathy of any cause, cardiac arrhythmias, or serious hepatic or renal disease
* Pregnancy or breast feeding
* Current use of medication with known serious hepatotoxic effects
* Current use of medication with known serious interaction with CQ: amiodarone, anticonvulsants, ciclosporin, digoxin, mefloquine, moxifloxacin
* Current severe depression (as indicated by current use of antidepressant medication)
* Known serious retinal disease
* Current or recent (within the past 30 days) participation in any other clinical intervention trial.
* Known G6PD deficiency
* Vaccination for influenza (seasonal or H1N1 strain) within the 3 months prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1516 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Laboratory-confirmed influenza-like illness | 12 weeks

SECONDARY OUTCOMES:
Serologically-confirmed influenza infection (symptomatic or asymptomatic) | 12 weeks
  Four-fold rise in influenza antibody titre at week 12 compared to the baseline sample

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas I Paton, MD FRCP, Study Chair — National University of Singapore; Lawrence Lee, MD PhD, Principal Investigator — National University of Singapore
Locations (1):
- Investigational Medicines Unit, National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Paton NI, Lee L, Xu Y, Ooi EE, Cheung YB, Archuleta S, Wong G, Wilder-Smith A. Chloroquine for influenza prevention: a randomised, double-blind, placebo controlled trial. Lancet Infect Dis. 2011 Sep;11(9):677-83. doi: 10.1016/S1473-3099(11)70065-2. Epub 2011 May 5. PMID 21550310